CLINICAL TRIAL: NCT00812058
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Study to Assess the Safety, Tolerability and Efficacy of RG2417 (Uridine) in the Treatment of Bipolar I Depression
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of RG2417 in Bipolar I Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Responsible Party: Hedy Dion, Repligen Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG2417-03
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar I Depression
Keywords: Bipolar Depression; Bipolar Disease; Bipolar Disorder; Bipolar; Manic Depression; Manic Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Uridine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RG2417 (Experimental): Oral RG2417 taken twice daily for 8 weeks
  Interventions: Drug: RG2417
- Placebo (Placebo Comparator): Oral placebo taken twice daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RG2417 — 1g bid dose escalates to 2g bid for weeks 2-8.
  Other Names: Uridine
  Arms: RG2417
Drug: Placebo — Similarly sized placebo pills to be taken in the same fashion as the RG2417 tablets.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to test a new drug, RG2417, to see how the drug affects symptoms of bipolar I depression and to make sure it is safe in humans.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I Disorder, most recent episode depressed
* History of 2 or more manic or mixed episodes, at least one of which required pharmacologic treatment for manic symptoms

Exclusion Criteria:

* Current manic, hypomanic or mixed episode
* Rapid cycling bipolar disorder (4 or more mood episodes in the last year)
* Dementia or any other Axis I diagnosis (besides bipolar I) that requires treatment
* Alcohol or drug dependence within 6 months; alcohol or drug abuse within 3 months
* Positive urine drug test for amphetamines, cocaine metabolites, opiates and/or phencyclidine(PCP)
* Axis II diagnosis likely to interfere with study compliance
* Serious suicidal or homicidal risk
* Sensitivity to any of the drug ingredients, including lactose
* Women who are pregnant, breast feeding or refuse to use adequate birth control
* Current seizure disorder
* Current episode of depression is longer than 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
MADRS Score | Baseline and weekly for 8 weeks

SECONDARY OUTCOMES:
CGI-BP-S | Baseline and weekly for 8 weeks
Safety Findings (includes AE frequency, YMRS Score and CSSR-S Score) | Baseline, 8 weeks of study drug dosing and one follow up visit at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sachs, MD, Principal Investigator — Massachusetts General Hospital
Locations (36):
- United States (36):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - K&S Professional Research Services, Little Rock, Arkansas
  - Affiliated Research Institute, San Diego, California
  - Yale University, New Haven, Connecticut
  - Behavioral Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solution, Inc., Orlando, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Valle Vista Health System, Greenwood, Indiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Department of Pscyhiatry & Psychology, Rochester, Minnesota
  - Behavioral Medical Research of States Island, Staten Island, New York
  - Unvieristy of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Richard H. Weisler, MD, PA and Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Western Psychiatric Institute Clinic, Pittsburgh, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - CNS Healthcare, Memphis, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - FutureSearch Trials of Austin, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - University of Texas, Houston Medical Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Dean Foundation, Middleton, Wisconsin